CLINICAL TRIAL: NCT00972751
Title: Investigation of Thioredoxin-1 Family Protein Expression in Rectal Cancer
Brief Title: S9304A Study of Protein Expression in Tumor Tissue Samples From Patients With Stage II or Stage III Rectal Cancer Enrolled in Clinical Trial SWOG-9304
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000601255; U10CA032102 (NIH); SWOG-9304A-ICSC (Other: SWOG)
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at protein expression in tumor tissue samples from patients with stage II or stage III rectal cancer enrolled in clinical trial SWOG-9304.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine expression levels of thioredoxin-1 (Trx-1), thioredoxin-interacting protein (TXNIP), and hypoxia inducible factor-1 alpha (HIF-1α) in paraffin-embedded resected tumor tissue samples from patients with stage II or III rectal cancer enrolled in clinical trial SWOG-9304.
* Determine if there is a correlation between Trx-1 and TXNIP expression and HIF-1α expression.
* Correlate expression of these proteins with tumor stage, disease-free survival, overall survival, and risk of recurrence.
* Determine interactions for patient age, performance status, and type of therapy received on clinical trial SWOG-9304.

OUTLINE: This is a multicenter study.

Paraffin-embedded resected tumor tissue samples are analyzed for protein expression levels (thioredoxin-1, thioredoxin-interacting protein, and hypoxia inducible factor-1 alpha) by tissue microarray and immunostaining.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Stage II or III disease
  * No metastases
* Enrolled on clinical trial SWOG-9304

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on SWOG-9304, adenocarcinoma of the recturm Stage II or III
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Expression of thioredoxin-1, thioredoxin-interacting protein, and hypoxia inducible factor-1 alpha | upon testing of specimens
Correlation of expression of these proteins with tumor stage, disease-free survival, overall survival, and risk of recurrence | upon provision of expression to Statistical Center

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Dragovich, MD, PhD, Study Chair — University of Arizona